CLINICAL TRIAL: NCT02331836
Title: Endocuff-assisted Versus Cap-assisted Versus Standard Colonoscopy for Adenoma Detection: A Randomized Controlled European Multicenter Study
Brief Title: Endocuff-assisted Versus Cap-assisted Versus Standard Colonoscopy
Acronym: EC-Cap-SC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Albert-Schweitzer-Klinik Northeim (Other)
Responsible Party: Principal Investigator, Tobias Meister, Prof. Dr. med. Tobias Meister, Helios Albert-Schweitzer-Klinik Northeim
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: EC-CUFF-2015
Record Dates: First submitted 2015-01-02; First posted 2015-01-06 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Polyps; Colorectal Adenomas
Keywords: adenoma detection rate; polyp detection rate; withdrawal time; coecal and ileum intubation rate
MeSH Terms: interventions — Contraceptive Devices, Female

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arc Endocuff (AEC 110, 120, 130, 140) (Active Comparator): Endocuff-assisted colonoscopy Colonoscopy with the Endocuff attached at the distal tip of the scope
  Interventions: Device: Arc Endocuff (AEC 110, 120, 130, 140)
- Cap (Active Comparator): Cap-assisted colonoscopy Colonoscopy with the transparent Cap attached at the distal tip of the scope
  Interventions: Device: Cap
- Standard Colonoscope (Active Comparator): Standard colonoscopy without any additional device
  Interventions: Device: Standard colonoscope

INTERVENTIONS:
Device: Arc Endocuff (AEC 110, 120, 130, 140)
  Arms: Arc Endocuff (AEC 110, 120, 130, 140)
Device: Cap — Olympus Disposable distal attachment 15mm diameter, 4mm depth
  Arms: Cap
Device: Standard colonoscope
  Arms: Standard Colonoscope

SUMMARY:
Comparison of Endocuff-assisted, Cap-assisted and Standard colonoscopy for assessment of the adenoma detection rate (ADR)

DETAILED DESCRIPTION:
The Endocuff is a medical device, approved in 2012 by the American Food and Drug Administration, which was also authorized by the European Agency for the Evaluation of Medicinal Products. The aim of the cuff is to optimize the view of the colonic mucosa. There is also a transparent cap on the market, which is used in colonoscopy for a better evaluation of the mucosa and polyp detection. The goal of this project is to conduct a prospective randomized trial for clarification of the hypotheses, whether the usage of the Endocuff increases the detection rate of adenomas compared to the transparent cap or compared to standard colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Colonoscopy independent from indication
* Age ≥ 18
* Patient is able to provide informed consent for the procedure

Exclusion Criteria:

* Inflammatory Bowel Disease stenosis
* Pregnant of nursing patient
* Acute diverticulitis
* Active Inflammatory Bowel Disease
* Age ≤ 18
* Coagulation disorder (INR>1.4 , Thrombocytes < 50000/µl)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | 1 year
  Proportion of patients having at least one adenoma
Polyp detection rate | 1 year
  Proportion of patients having at least one adenoma

SECONDARY OUTCOMES:
Bowel preparation result | one day
Coecum intubation rate | one year
Ileum intubation rate | one year
Coecum intubation time | one day
withdrawal time | one day
mucosal laceration | one day
severe bleeding | one day
perforation | one day

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Meister, Prof. Dr.med., Principal Investigator — Helios Albert-Schweitzer-Hospital
Locations (6):
- Germany (5):
  - University of Muenster, Münster, North Rhine-Westphalia
  - University Medical Center Göttingen, Göttingen
  - HELIOS St. Marienberg Klinik Helmstedt, Helmstedt
  - HELIOS Albert-Schweitzer-Klinik, Northeim
  - HELIOS Medical Center Siegburg, Siegburg
- Wroclaw Medical University, Wroclaw, Poland